CLINICAL TRIAL: NCT01869439
Title: Utilizing Visual and Thermal Images for the Measuring and Monitoring of External Wounds
Brief Title: Measuring Wounds Found on the Outside of the Body Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wound Vision (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WV12CL-0003 Revision 09
Record Dates: First submitted 2013-05-22; First posted 2013-06-05 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: External Wounds Measured for Length by Width Using a Ruler
Keywords: Pressure Ulcers; Bed Sores; Measuring; Visual Images; Thermal Images; External Wounds; Area; Length; Width; Gradient
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- External wounds measured for length by width using a ruler (Experimental): This is a single arm study of subjects who have an external wound that is currently measured for length and width using a ruler. A study subject may have up to 3 qualifying external wounds.
  Interventions: Device: "gold standard" LxW manual ruler measurement technique; Device: WMMS ImageReview software's LxW measurement technique; Device: WMMS ImageReview software's Visual External Wound Trace; Device: WMMS ImageReview software's External Wound Trace Overlay

INTERVENTIONS:
Device: "gold standard" LxW manual ruler measurement technique — Currently, the "gold standard" LxW manual ruler measurement technique is used for measuring the area of an external wound. The LxW is measured by measuring the longest length (head to toe) times the widest width (perpendicular to the length).
Device: WMMS ImageReview software's LxW measurement technique — This software measurement technique is part of tthe WMMS and also measures the external wound LxW by the longest length (head to toe) times the widest width (perpendicular to the longest length).
Device: WMMS ImageReview software's Visual External Wound Trace — This is a measurement technique of the ImageReview software that enables the user to trace the perimeter edge of the wound's visual image.
Device: WMMS ImageReview software's External Wound Trace Overlay — This measurement technique is a feature of the WMMS, utilizing the visual external wound trace and overlaying it onto the thermal wound site. From the thermal overlay, variation data such as the differences in the thermal intensities (gradient), mean, and the mode of the thermal wound bed can be measured.

SUMMARY:
The purpose of this study is to test wounds found on the outside of the body surface with an investigational medical imaging device that collects visual pictures and thermal digital pictures of the wound site. The investigational device has not been approved by the Food and Drug Administration (FDA).

The medical imaging device is non-contacting and is non-radiating (delivers no energy to the body). It passively collects pictures (typical digital color photographs)and thermal pictures (black and white digital photographs of heat at the body surface.)

DETAILED DESCRIPTION:
This prospective study utilizes the WoundVision Wound Measuring and Monitoring System (WMMS) to study external wounds, which can currently be measured for length by width using a ruler. WMMS operates by taking simultaneous visual and thermal images of the external wound site and the associated body surface. These images are evaluated by utilizing the WMMS ImageReview measuring and monitoring software. WMMS ImageReview software allows for LxW (length by width) and surface area (cm squared),as well as perimeter (cm) external wound measurements of the visual image. WMMS ImageReview software also allows for the display of thermal intensity variation data for the associated body surface of the corresponding thermal image.

This study is primarily designed to utilize the Coefficients of Individual Agreement (CIA)as a means of establishing the equivalence of area measurements utilizing the WMMS ImageReview software LxW technique and the current "gold standard" LxW manual ruler technique.

A secondary objective measures the thermal intensity variation data of the external wound bed by overlaying the corresponding "Visual External Wound Trace"from the visual image onto the thermal wound bed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater, of either gender and of any ethnic background
* Able to tolerate position changes and turns for up to 10 minutes comfortably
* Have an existing external wound that is currently measured for length and width using a ruler

  * The protocol will allow imaging up to 3 external wounds per subject
  * The 3 external wounds must be in separate body locations (ex: one on the right heel, one on the left heel, and the other on the sacrum).
* Have qualifying external wound sites:

  * External wounds whose external wound site fits entirely within the field of view and do not wrap around a body edge.
  * No device or treatment will obscure the external wound site

Exclusion Criteria:

* Neonatal and pediatric patients
* Pregnant women
* Cannot tolerate position changes for up to 10 minutes comfortably (per external wound site imaged)
* Cannot be positioned so images can be taken at approximately 90 degrees perpendicular and 18 inches away from the external wound site
* On therapies or treatments which cannot be safely suspended long enough to conduct an imaging session as determined by facility policy
* Have external wound dressing or medical device which cannot or should not be removed as determined by site investigator
* Have an external wound with excessive or heavy exudate that cannot be controlled during the imaging session. Excessive drainage can obscure external wound features
* Have complex external wound site(s):

  * The external wound wraps around a body edge or otherwise cannot be imaged entirely within the visual field of view
  * From visual assessment the existing external wound cannot be clearly distinguished from other conditions at the external wound site (e.g. break down or the deterioration of the surrounding body surfaces due to other conditions such as cancer or other types of wounds makes determining the edge of the external wound impossible)
* Have not provided signed informed consent
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: V. Chowdry Pinnamaneni, M.D., Principal Investigator — St.Vincent Wound Healing Center
Locations (2):
- United States (2):
  - St. Vincent Seton Specialty Hospital, Indianapolis, Indiana
  - St. Vincent Wound Healing Center, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Wounds Measures of LxW Ruler & Software LxW, Area & Perimeter: This is a single arm study of subjects who have an external wound that is currently measured for length and width using a ruler. A study subject may have up to 3 qualifying external wounds.
  "gold standard" LxW manual ruler measurement technique: Currently, the "gold standard" LxW manual ruler measurement technique is used for measuring the area of an external wound. The LxW is measured by measuring the longest length (head to toe) times the widest width (perpendicular to the length).
  WMMS ImageReview software's LxW measurement technique: This software measurement technique is part of tthe WMMS and also measures the external wound LxW by the longest length (head to toe) times the widest width (perpendicular to the longest length).
  WMMS ImageReview software's Visual External Wound Trace: This is a measurement technique of the ImageReview software that enables the user to trace the perimeter edge of the wound's visual image.
Period: Overall Study
Arm/Group | Wounds Measures of LxW Ruler & Software LxW, Area & Perimeter
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- External Wounds Measured for Length by Width Using a Ruler: This is a single arm study of subjects who have an external wound that is currently measured for length and width using a ruler. A study subject may have up to 3 qualifying external wounds.
  "gold standard" LxW manual ruler measurement technique: The LxW is measured by measuring the longest length (head to toe) times the widest width (perpendicular to the length).
  LxW measurement technique: This software measurement technique measures the external wound LxW by the longest length (head to toe) times the widest width (perpendicular to the longest length).
  Visual External Wound Trace: This software measurement enables the user to trace the perimeter edge of the wound's visual image.
  External Wound Trace Overlay: This software measurement utilizes the visual external wound trace and overlaying it onto the thermal wound site. From the thermal overlay, data such as the differences in the thermal intensities (gradiency), mean, and the mode of the thermal wound bed can be measured.
Arm/Group | External Wounds Measured for Length by Width Using a Ruler
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  >18 years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Within and Between Reader Agreement for the Measurement Techniques: Scout Length by Width, Scout Trace Area, and Scout Trace Perimeter
Description: Establish within and between reader agreement of the Scout Length by Width, Scout trace area, and Scout trace perimeter.
Time Frame: 90 Days
Population: 40 wounds captured in an inpatient and outpatient population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of CV
Groups:
- Wounds Measured for Length by Width Using a Ruler and Software: This is a single arm study of subjects who have an external wound that is currently measured for length and width using a ruler. A study subject may have up to 3 qualifying external wounds.
  The "gold standard" LxW manual ruler measurement technique: Currently, the "gold standard" LxW manual ruler measurement technique is used for measuring the area of an external wound. The LxW is measured by measuring the longest length (head to toe) times the widest width (perpendicular to the length).
  Software LxW measurement technique: This software measurement technique is part of tthe WMMS and also measures the external wound LxW by the longest length (head to toe) times the widest width (perpendicular to the longest length).
  Software's Visual External Wound Trace: This is a measurement technique of the ImageReview software that enables the user to trace the perimeter edge of the wound's visual image.
Arm/Group | Wounds Measured for Length by Width Using a Ruler and Software
Number analyzed (Participants) | 40
percentage of CV
  Between Reader Software LxW Area | 20.07 (16.71)
  Between Reader Software Trace Area | 16.28 (16.10)
  Between Reader Software Perimeter | 16.28 (5.82)
  Within Reader Software Trace Area | 20.07 (8.68)
  Within Reader Area by Software Measurement | 16.28 (6.46)
  Within Reader Software Perimeter | 16.28 (3.32)

ADVERSE EVENTS:
Arm/Group | External Wounds Measured for Length by Width Using a Ruler
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less